CLINICAL TRIAL: NCT02657824
Title: Rapid and Easy Evaluation of Cardiac Systolic Function by Means of Mitral Valve Movements in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Neslihan Siliv, doctor, Bozyaka Training and Research Hospital
Other Study IDs: 06072015
Record Dates: First submitted 2015-12-22; First posted 2016-01-18 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-01

CONDITIONS: Heart; Disease, Mitral(Valve)
Keywords: Ejection fraction; mitral valve; e-point septal separation
MeSH Terms: conditions — Disease

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- measuring ejection fraction: ejection fraction in an acute dyspneic patients
  Interventions: Other: dyspneic patients

INTERVENTIONS:
Other: dyspneic patients — measuring mitral valve and septal distance in acute dyspneic patients for estimating left ventricular ejection fraction

SUMMARY:
Left ventricular ejection fraction (LVEF) is a parameter that should be evaluated rapidly to the patients, admitted to the emergency department with shortness of breath. The investigators aimed to investigate correlation between LVEF and 4 different mitral valve movements which alternate to the classical LVEF assessing methods and evaluate these methods can be used or not in the emergency department.

DETAILED DESCRIPTION:
A prospective observational study was conducted in an acutely dyspneic patients with receiving echocardiagraphy by the chief physicians. Measurements were performed before echocardiography lab by the physician who conducted the survey in the emergency department. In parasternal long axis view mitral valve E-Point Septal Separation (EPSS) M-Mod measurements and mitral valve anterior leaflet and septal distance (P-ALSS) B-Mod measurements and in apical four chamber view mitral valve anterior leaflet and septal distance (A-ALSS) B-Mod measurements and distance between mitral valve anterior and posterior leaflets (MVLS) B-Mod measurements were acquired as the minimum distance in diastole. LVEF of patients were measured by cardiologist. Correlation of the all values between LVEF and sensitivity, specificity, and likelihood probabilities were calculated.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* nontraumatic acute dyspneic patients

Exclusion Criteria:

* sigmoid septum
* septal hypertrophia
* mitral stenosis
* mitral valve prothesis
* aortic regurgitation
* regional wall motion defect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: an acutely dyspneic patients with receiving echocardigraphy by the chief physicians in the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2015-08; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Dyspneic patients were evaluated for their left ventricular ejection fraction by new methods with using transthoracic echocardiography. | up to 2 hours after admitting to the emergency department
  New methods are described: First measurement is distance between mitral valve anterior leaflet and septum in early diastole in the parasternal long axis view m-mode in millimeter.second measurement is distance between mitral valve anterior leaflet and septum in early diastole in the parasternal long axis view b-mode in millimeter. third is the distance between mitral valve anterior leaflet and septum in the apical four chamber view b-mode in millimeter. forth is the distance between mitral valve anterior and posterior leaflet in apical four chamber b-mode in millimeter.

CONTACTS AND LOCATIONS:
Overall Officials: neslihan siliv, Principal Investigator — ızmır bozyaka traınıng and research hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Secko MA, Lazar JM, Salciccioli LA, Stone MB. Can junior emergency physicians use E-point septal separation to accurately estimate left ventricular function in acutely dyspneic patients? Acad Emerg Med. 2011 Nov;18(11):1223-6. doi: 10.1111/j.1553-2712.2011.01196.x. Epub 2011 Nov 1. PMID 22044429
- [Result] Weekes AJ, Reddy A, Lewis MR, Norton HJ. E-point septal separation compared to fractional shortening measurements of systolic function in emergency department patients: prospective randomized study. J Ultrasound Med. 2012 Dec;31(12):1891-7. doi: 10.7863/jum.2012.31.12.1891. PMID 23197541
- [Result] McKaigney CJ, Krantz MJ, La Rocque CL, Hurst ND, Buchanan MS, Kendall JL. E-point septal separation: a bedside tool for emergency physician assessment of left ventricular ejection fraction. Am J Emerg Med. 2014 Jun;32(6):493-7. doi: 10.1016/j.ajem.2014.01.045. Epub 2014 Feb 3. PMID 24630604